CLINICAL TRIAL: NCT01416883
Title: Oral Mucosal Absorption Study of ICI176,334-1 (Bicalutamide New Formulation) in Japanese Healthy Male Subjects
Brief Title: Oral Mucosal Absorption Study of Bicalutamide New Formulation
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Gerard Lynch, AstraZeneca
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D6874L00016
Record Dates: First submitted 2011-08-12; First posted 2011-08-15 (Estimated); Last update posted 2011-08-15 (Estimated); Status verified 2011-08

CONDITIONS: Healthy
Keywords: oral mucosal absorption; pharmacokinetics; safety; bicalutamide; Japanese; healthy subject

ARMS (1):
- Active 1 (Experimental): 8 subjects will receive ICI176,334-1
  Interventions: Drug: ICI176,334-1

INTERVENTIONS:
Drug: ICI176,334-1 — Subject will receive single dose of ICI176,334-1

SUMMARY:
The purpose of this study is to investigate the presence or absence of oral mucosal absorption of bicalutamide after ICI176,334.1 is given to Japanese healthy male subjects

DETAILED DESCRIPTION:
Oral mucosal absorption study of ICI176,334-1 (Bicalutamide new formulation) in Japanese healthy male subjects

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent prior to any study specific procedures
* Japanese healthy male subjects aged 20 to 45 years
* Male subjects should be willing to use barrier contraception ie, condoms, until 3 months after the last dose of investigational product
* Have a body mass index (BMI) between 17 and 27 kg/m2
* Eligible based on the physical findings, supine BP, pulse rate, ECG and laboratory assessments, as judged by the investigator(s)

Exclusion Criteria:

* Presence of any disease under medical treatment
* History or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, immunological, blood, endocrine, neurological or mental disease to interfere with absorption, distribution, metabolism or excretion of drugs judged by investigator(s)
* Presence of any infectious disease, such as bacteria, virus and fungus Presence of allergic disorder, such as asthma, pollen disease or atopic dermatitis, and judged as necessary any medical treatment
* Any large surgical history of gastrointestinal tract such as gastric/intestinal resection or suturation

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2010-07; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
To investigate the presence or absence of oral mucosal absorption of ICI176,334-1 by assessment of concentration of bicalutamide in saliva. | Blood samples are taken repeatedly for 72 hours and also taken at 168 hours after application of the investigational drug.
To investigate the presence or absence of oral mucosal absorption of ICI176,334-1 by assessment of concentration of bicalutamide in plasma. | Blood samples are taken repeatedly for 72 hours and also taken at 168 hours after application of the investigational drug.

SECONDARY OUTCOMES:
To assess the safety by assessment of adverse event. | Subjects will be monitored for adverse events prior to treatment and up to 14 to 21 days (follow-up) after application of the investigational drug.
To assess the safety by assessment of vital signs. | Subjects will be monitored for vital signs prior to treatment and up to 14 to 21 days (follow-up) after application of the investigational drug.
To assess the safety by assessment of electrocardiograms (ECGs). | Subjects will be monitored for electrocardiograms (ECGs) prior to treatment and up to 14 to 21 days (follow-up) after application of the investigational drug.